CLINICAL TRIAL: NCT01098214
Title: The Role of Cytokines (and Other Biomarkers) in Apparently Normal Pregnancies
Brief Title: The Role of Cytokines in Apparently Normal Pregnancies
Status: Withdrawn | Type: Observational
Why Stopped: Decided not to pursue study at this time. Resources not available
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 09310
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Pregnancy
Keywords: Normal pregnancy; Amniotic fluid; Cytokines; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Amniotic fluid samples from patients undergoing amniocentesis with an apparently normal pregnancy will have a small aliquot of fluid stored for future analysis, including the cytokine profile, proteomics, metabolomics, etc.
Oversight: Data Monitoring Committee: No

SUMMARY:
To provide rigorous, detailed normative data for diagnostics and comparative studies, to determine relationships between cytokine levels (and other biomarkers) and clinical data, and gain further insight into the pro-/anti-inflammatory cytokine profile of normal midtrimester amniotic fluid.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Pregnancies between 15-25 weeks gestation.
* Able to provide informed consent.
* No apparent major sonographic abnormality.

Exclusion Criteria:

* Any major fetal anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing amniocentesis with an apparently normal pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazeeh Hanna, M.D., Principal Investigator — Winthrop University Hospital